CLINICAL TRIAL: NCT04930523
Title: Effect of Spinal Decompression With and Without ELDOA in Patients of Lumber Disc Protrusion
Brief Title: Effect of Decompression With and Without ELDOA in Lumber Disc Protrusion Patients
Acronym: ELDOA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aqua Medical Services (Pvt) Ltd (Industry)
Responsible Party: Principal Investigator, Mir Arif Hussain, Research Head, Aqua Medical Services (Pvt) Ltd
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Kenza Rehman 00379
Record Dates: First submitted 2021-06-11; First posted 2021-06-18 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Lumbar Disc Herniation
Keywords: ELDOA; Disc herniation; Decompression; LBP
MeSH Terms: conditions — Intervertebral Disc Displacement | interventions — Decompression

STUDY DESIGN:
Intervention Model Description: Control group will be treated by decompression session while experimental group will be treated with ELDOA along with decompression.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decompression (Active Comparator): It include the pre- Physiotherapy treatment than decompression and post physiotherapy treatment.
  Interventions: Other: Decompression
- Experimental (Experimental): It includes the Pre physiotherapy treatment than ELDOA positions are guided and performed by patients before decompression Low back exercises guided i.e. knee to chest, pelvic rolling, bridging, SLR, piriformis exercises is guided for home plan along with precaution and Decoarctation of (C0/C1/C2),(C4/C5),(C5,C6),(C6/C7),(T4/T5),(T6/T7),(T8,/T9),(L4/L5),(L5/S1) then Neuro-oxy motorized lumbar spinal decompression therapy for 25 minutes and at last Post physiotherapy treatment
  Interventions: Other: Elongation Longitudinaux Avec Decoaption Osteo Articulaire

INTERVENTIONS:
Other: Elongation Longitudinaux Avec Decoaption Osteo Articulaire — Pre physiotherapy treatment
  Gym (treadmill ,cycling,vibrator) according to ability and condition of patient Shortwave diathermy SWD for atleast 10 mins Decompression treatment i.e. Neuro-oxy motorized lumbar spinal decompression therapy for 25 minutes.
  Post physiotherapy treatment
  Conventional Tens and infrared heat for 10 minutes at low back region. TENS is modality to reduce pain and tension,by stimulating large diameter afferent fiber .IR give superficial heat for circulation and relaxation of muscles.
  No exercises or walk were guided for home (till 24 hrs) Low back exs guided i.e knee to chest, pelvic rolling, bridging, SLR, pirformis exs is guided for home plan along with precautions.
  No exertion ,drive carefully Avoid stairs climbing ,twisting ,bending ,weight lifting
  Arms: Experimental
Other: Decompression — Pre physiotherapy treatment
  Gym (treadmill ,cycling, vibrator) according to ability and condition of patient Shortwave diathermy SWD for at least 10 minutes. ELDOA positions are guided and performed by patients before decompression Low back exercises guided i.e. knee to chest, pelvic rolling, bridging, SLR, piriformis exercises is guided for home plan along with precautions.
  Decoarctation of (C0/C1/C2),(C4/C5),(C5,C6),(C6/C7),(T4/T5),(T6/T7),(T8,/T9),(L4/L5),(L5/S1) Neuro-oxy motorized lumbar spinal decompression therapy for 25 minutes. Post physiotherapy treatment Tens and infrared heat for 10 minutes at low back region. TENS is modality to reduce pain and tension, by stimulating large diameter afferent fiber .IR give superficial heat for circulation and relaxation of muscles.
  ELDOA exercises(positions)are guided for home plan after session (after 24 hrs) No exertion ,drive carefully Avoid stairs climbing, twisting bending, weight lifting
  Arms: Decompression

SUMMARY:
The study will be conducted to determine the effects of spinal decompression with and without ELDOA in patients of lumbar disc protrusion. A total of twenty patient with lumber disc protrusion will be taken after fulfilling the inclusion criteria. the patient will be divided in experimental group i.e. ELDOA along with decompression and control group. Both session got pre and post session along with general low back exs.home plan along with precautions was guided to every patient of control and experimental group.NPRS ,ODI is assess in first and fourth session. The data will be analyzed through IBM SPSS version 21.

DETAILED DESCRIPTION:
Low back pain due to lumber disc protrusion is common health problem in all population, which affects the normal activities of daily living by decreasing the functional status due to low back pain that rad to leg. Literature supports that decompression have significant effect in improving the functional status of patient with low back pain with radiation but reoccurrence of problem of this problem is common with this problem. So my study is aiming to find the effectiveness of ELDOA along with decompression to minimize the re occurrence of low back and functional status. ELDOA will help to tone up the fascia and strengthen the spinal muscles The intervertebral disc consists of an inner nucleus pulposus (NP) and an outer annulus fibroses (AF). The central NP area which facilitate water retention, creating hydrostatic pressure to resist axial compression of the spine. The NP is primarily composed of type II collagen, which accounts for 20% of its overall dry weight. In contrast, the AF functions to maintain the NP within the center of the disc with low amount of PG; 70% of its dry weight is comprised of primarily concentric type I collagen fibers . In LDH, narrowing of the space available for the thecal sac can be due to protrusion of disc through an intact AF, extrusion of the NP through the AF though still maintaining continuity with the disc space, or complete loss of continuity with the disc space and sequestration of a free fragment.

Motorized table with mechanical space in between two parts of table. Pelvic and thoracic belt is tie at lumber and thoracic level to fasten the patient. Static, intermittent and cycling distractive force applied to lumber area for minute. Distraction(angle of pull) and relaxation force is monitored by therapist. Specific disc that cause pain and other symptoms are targeted .curves on computer help to reduce muscle spasm. Antigravity force applied on lumber area in the space and pull backward protrude disc. Biofeedback computer module in which number of session depends upon medical condition age .targeted level of spine is selected. neuro oxy spinal decompression non-surgical and cost effective Treatment that stimulate natural healing of injured and degenerative vertebra. Works on decompressing and lengthening the spine with chronic pains. These movement produce negative pressure in the disc as a result vacuum created as a result bulge, protrude part repositioned and align. Nourishment of injured area is restore by oxygen and nutrients. Pressure on nerve relives patient feel symptoms free. Special senses in machine that detect limitation and tension of patient results of spinal decompression is better than traditional traction. Other name of decompression is intervertebral differential dynamic therapy, mechanical spinal distraction therapy. Negative pressure is created between vertebras so that protruded part pull inward and nerve become free from pressure. Table has two parts which is separated with space where distractive force apply on spine. Two belts thoracic and lumber to fasten the patient. Pulling force is minimal last for a minute depend upon patient symptoms can be adjusted to static, intermittent and cycling control by therapist to induce relaxation. During treatment antigravity force applied at spine automatically by machine system and helps to move protruded part back to position as a result nerve get pressure free. Treatment is painless, gentle and intermittent.

Guy voyer is the founder of Elongation longitudinaux avec decoaption osteoarticulaire or LOADS longitudinal osteo articular decoaptation stretching .This exercise specifically work on every spinal level. Fascial stretch along with tension at spinal level. Strength of the back muscles and stretching of paraspinal work to improve the tone. Concept is based that micro movement affects macro movement as a result function betters. Spine contains 24 segments c0/c1/c3 and end to L5/S1.Fascia attach to vertebral bodies anteriorly. Posteriorly osseous framework ,muscles attach with bones ,bony framework include zygapophyseal joints that guide movements , ligament structure restrict the movement.Disc that is sponge act as shock absorption. Neurological and circulatory system work to continue functioning. They effect body locally and generally. Local effects in reducing degeneration by mobilizing the zygapophyseal joints exchange of fluid with absorption, improve arterial and venous circulation that help to remove waste and improve circulation, improve tone ROM ,posture and alignment.

General effects include postural correction by supporting systems ,limbs ,muscles. Improve respiratory mechanism that restore the flow of CSF,effect psychosomatic component make balance between mind and body,neurohormonal facilitation by improving autonomic function improvement and proper functioning,propioreception improvement by self-correcting poor posture, fascia work in coordinated chain manner and help to decrease the energy consumption.

ELIGIBILITY:
Inclusion Criteria:

* Both Gender
* Age b/w 25 to 65
* Limited ROM
* Pain more than 3 on NPRS

Exclusion Criteria:

* Malignancy.
* Infection.
* Trauma.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2021-07-11 (Actual); Study Completion 2021-07-20 (Actual)

PRIMARY OUTCOMES:
Numeric pain rating scale | 4th weeks
  It is numeric pain rating scale for measuring pain intensity. it ranges from 0-10.In which 0 shows no pain,1-3 (mild pain),4-6(moderate pain) and 10 shows severe pain. As guided by the researcher, pain intensity was marked by the patient
Oswestry Disability Index (ODI) | 4th weeks
  Oswestry disability index is important tool in spinal disorders patients. Disability is measured by questioner related to activities of daily living. This tool is use for every type of patient acute or chronic with severe spinal disability. Each question contain 6 items from 0 to 5 i.e. no pain, mild , moderate, severe, very severe, worst.0 to 20 is minimal disability,21 to 40 is moderate,41 to 60 is severe,61 to 80 is crippled and 81 to 100 bed bound patient
Inclinometer | 4th week
  Inclinometer is an instrument to measure range of motion or angle of motion of spine. Two inclinometer is use to measure dynamic motion of spine. There is motion on both ends of spine .in order to find true angle One inclinometer is on upper spine and other is on lower spine and value of lower spine is subtracted from upper spine.
  The flexion,, extension and side bending towards the right and left will be checked.

CONTACTS AND LOCATIONS:
Overall Officials: Kanza Rehman, MS-OMPT, Principal Investigator — Riphah International University
Locations (1):
- KKT Canada Orthopedic & Rehabilitation Centre, Rawalpindi, Capital, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheung KM, Karppinen J, Chan D, Ho DW, Song YQ, Sham P, Cheah KS, Leong JC, Luk KD. Prevalence and pattern of lumbar magnetic resonance imaging changes in a population study of one thousand forty-three individuals. Spine (Phila Pa 1976). 2009 Apr 20;34(9):934-40. doi: 10.1097/BRS.0b013e3181a01b3f. PMID 19532001
- [Background] Battie MC, Videman T, Parent E. Lumbar disc degeneration: epidemiology and genetic influences. Spine (Phila Pa 1976). 2004 Dec 1;29(23):2679-90. doi: 10.1097/01.brs.0000146457.83240.eb. PMID 15564917
- [Background] Luoma K, Riihimaki H, Luukkonen R, Raininko R, Viikari-Juntura E, Lamminen A. Low back pain in relation to lumbar disc degeneration. Spine (Phila Pa 1976). 2000 Feb 15;25(4):487-92. doi: 10.1097/00007632-200002150-00016. PMID 10707396
- [Background] Lee Y, Lee C-R, Cho M. Effect of decompression therapy combined with joint mobilization on patients with lumbar herniated nucleus pulposus. Journal of Physical Therapy Science. 2012;24(9):829-32.
- [Background] Rathod AK, Dhake RP. Radiographic Incidence of Lumbar Spinal Instability in Patients with Non-spondylolisthetic Low Backache. Cureus. 2018 Apr 4;10(4):e2420. doi: 10.7759/cureus.2420. PMID 29872600
- [Background] Waqqar S, Shakil-Ur-Rehman S, Ahmad S. McKenzie treatment versus mulligan sustained natural apophyseal glides for chronic mechanical low back pain. Pak J Med Sci. 2016 Mar-Apr;32(2):476-9. doi: 10.12669/pjms.322.9127. PMID 27182265
- [Background] Choi J, Lee S, Hwangbo G. Influences of spinal decompression therapy and general traction therapy on the pain, disability, and straight leg raising of patients with intervertebral disc herniation. J Phys Ther Sci. 2015 Feb;27(2):481-3. doi: 10.1589/jpts.27.481. Epub 2015 Feb 17. PMID 25729196
- [Background] Apfel CC, Cakmakkaya OS, Martin W, Richmond C, Macario A, George E, Schaefer M, Pergolizzi JV. Restoration of disk height through non-surgical spinal decompression is associated with decreased discogenic low back pain: a retrospective cohort study. BMC Musculoskelet Disord. 2010 Jul 8;11:155. doi: 10.1186/1471-2474-11-155. PMID 20615252